CLINICAL TRIAL: NCT04405778
Title: An Open-Label, Dose Escalation, Phase 1, First-in-Human Study of TAK-102 in Adult Patients With GPC3-Expressing Previously Treated Solid Tumors
Brief Title: A Study of TAK-102 in Adult With Previously-Treated Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision unrelated to patient safety
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAK-102-1501; U1111-1247-6429 (Other: WHO); jRCT1080225204 (Registry Identifier: jRCT)
Record Dates: First submitted 2020-05-26; First posted 2020-05-28 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TAK-102 Cohort 1 (Experimental): TAK-102, 1 × 10^7 Chimeric antigen receptor (CAR) (+) cells/body as a starting dose, intravenous infusion, will be administered at approximately 5 mL/min and completed within 60 minutes.
  Interventions: Biological: TAK-102
- TAK-102 Cohort 2 (Experimental): TAK-102, 1 × 10^8 CAR (+) cells/body as a starting dose, intravenous infusion, will be administered at approximately 5 mL/min and completed within 60 minutes.
  Interventions: Biological: TAK-102
- TAK-102 Cohort 3 (Experimental): TAK-102, 1 × 10^9 CAR (+) cells/body as a starting dose, intravenous infusion, will be administered at approximately 5 mL/min and completed within 60 minutes.
  Interventions: Biological: TAK-102

INTERVENTIONS:
Biological: TAK-102 — TAK-102 intravenous infusion

SUMMARY:
Some solid tumors make a lot of a protein called glypican 3(GPC3), which helps it to grow. Healthy cells and tissues do not make GPC3. TAK-102 is a medicine that sticks to GCP3 and stops it from working. It is hoped that TAK-102 will eventually treat people with solid tumors with the GPC3 protein. TAK-102 will be added to each person's white blood cells so is custom-made for each person.

In this study, people with solid tumors with GPC3 will receive TAK-102 with their white blood cells. The main aims of this study are to check if the participants get any side effects from treatment with TAK-102 and to check how much TAK-102 they can receive without getting side effects from it. Researchers can then work out the best dose of TAK-102 to give to participants in future studies.

At the first visit, the study doctor will check who can take part. For those who can take part, the study doctors will collect white blood cells from each participant. These cells are sent to the laboratory where TAK-102 is added to each participant's cells. This can take up to 4 weeks. Participants will receive specific treatments while they are waiting for TAK-102. Then, participants will receive TAK-102 with their cells slowly through a vein (infusion). 3 different small groups of participants will receive lower to higher doses of TAK-102. Each participant will just receive 1 dose. The study doctors will check for side effects after each different dose of TAK 102. In this way, researchers can work out the best dose of TAK-102 to give to participants in future studies.

Participants will stay in hospital for 28 days or longer for their treatment. Then, they will visit the clinic for regular check-ups for up to 36 months.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-102. TAK-102 is being tested to treat people who have GPC3-expressing previously treated solid tumors. This study will look at the safety and tolerability of TAK-102 and will determine the RP2D of TAK-102.

The study will enroll approximately 14 participants, with a maximum of 18 participants. Participants will be assigned to 1 of the 3 treatment groups (dose cohorts) and dose escalation will be conducted in this study:

* Cohort 1: 1 × 10^7 CAR (+) cells/body [starting dose].
* Cohort 2: 1 × 10^8 CAR (+) cells/body.
* Cohort 3: 1 × 10^9 CAR (+) cells/body.

In case Cohort 1 is not tolerable, the dose level will be de-escalated to Cohort -1: 3 × 10^6 CAR (+) cells/body. Dose level(s) between planned cohorts and/or other dosing schedules may also be tested.

This study consists of the Screening, Pretreatment, and Treatment and Primary Follow-up phases. In Treatment and Primary Follow-up phases, all participants will be asked to receive a single intravenous infusion of TAK-102 and administration of TAK-102 will continue up to Month 12.

This multi-center trial will be conducted in Japan. The overall time to participate in this study is up to 15 years (In general, the 12-month Treatment and Primary Follow-up, 2-year Secondary Follow-up and then 12-year Long Term Follow-up phases in another study). Participants will make multiple visits to the clinic and be hospitalized for at least 28 days to receive treatment with TAK-102 followed by a recovery period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged ≥18 years at the time of signing informed consent.
2. Participants must have a diagnosis of solid tumors.
3. Participants with solid tumor who are refractory or intolerant to standard treatments.
4. GPC3-expression must be determined on the tumor locally by IHC using a validated assay, scoring and staining confirmed by the sponsor prior to leukapheresis procedures.
5. Life expectancy ≥12 weeks.
6. ECOG performance status of 0 or 1.
7. Adequate organ function as confirmed by clinical laboratory values as specified below:

   1. Total bilirubin must be <1.5 × the upper limit of the normal range (ULN). Total bilirubin may be elevated up to 3 × ULN if the elevation can be reasonably ascribed to the presence of metastatic disease in the liver.
   2. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) must be <3 × ULN. AST and ALT may be elevated up to 5 × ULN if the elevation can be reasonably ascribed to the presence of metastatic disease in liver.
   3. Calculated creatinine clearance >50 mL/mins (The Cockcroft-Gault formula).
   4. Hemoglobin must be ≥8 g/dL.
   5. Neutrophil count must be >1000/mm^3.
   6. Absolute lymphocyte count must be >500/mm^3.
   7. Platelet count must be >75,000/mm^3.
   8. Prothrombin time-international normalized ratio must be ≤1.7.
   9. Activated partial thromboplastin time (APTT) must be ≤1.5 × ULN.
8. Participants must have radiographically measurable disease as defined by RECIST 1.1.
9. Female participants who:

   1. Are postmenopausal (natural amenorrhea and not due to other medical reasons) for at least 1 year before the screening visit, OR
   2. Are surgically sterile, OR
   3. If they are of childbearing potential, agree to practice 1 highly effective nonhormonal method of contraception and 1 additional effective (barrier) method at the same time, from the time of signing the informed consent through at least 12 months following TAK-102 infusion, OR
   4. Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant.

   Note: Periodic abstinence (eg, calendar, ovulation, symptothermal, postovulation methods), withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception.
10. Male participants, even if surgically sterilized (ie, postvasectomy), who:

    1. Agree to practice effective barrier contraception from the time of signing the informed consent through at least 12 months following TAK-102 infusion, OR
    2. Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant.

    Note: Periodic abstinence (eg, calendar, ovulation, symptothermal, postovulation methods), withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception.
11. Voluntary written consent must be given before performance of any study-related procedures not part of standard medical care, with the understanding that consent may be withdrawn by the participant at any time without prejudice to future medical care.
12. Willingness and ability to comply with scheduled visits and study procedures.

Exclusion Criteria:

1. Active systemic infections excluding well-controlled chronic HBV/HCV infections, coagulation disorders, or other major medical illnesses including cardiovascular, respiratory or immune system, myocardial infarction, cardiac arrhythmias, and obstructive/restrictive pulmonary disease.
2. Participants with known cardiopulmonary disease defined as unstable angina, clinically significant arrhythmia, congestive heart failure. A well-controlled atrial fibrillation would not be an exclusion whereas uncontrolled atrial fibrillation would be an exclusion.
3. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
4. Patients with any signs of lymphoma and/or leukemia
5. Patients who are diagnosed with or treated for another malignancy within 3 years before leukapheresis procedures. Patients with nonmelanoma skin cancer or carcinoma in situ (eg, cervix, bladder, breast) would be included if they were adequately treated.
6. Active, serious infection requiring antibiotics.
7. Any disease requiring systemic steroid treatment or steroid inhalant.
8. Any prior use of cell and gene therapy(ies).
9. Treatment with any investigational products (except for cell or gene therapy) within 14 days before leukapheresis procedures or 28 days before treatment with preconditioning chemotherapy/TAK-102.
10. Systemic anticancer therapy (including platinum-based chemotherapies and I/O therapies) within 14 days before leukapheresis procedures or treatment with preconditioning chemotherapy/TAK-102.
11. Treatment with radiotherapy within 14 days before leukapheresis procedures or treatment with preconditioning chemotherapy/TAK-102.
12. Treatment with major surgery within 28 days before leukapheresis procedures or treatment with preconditioning chemotherapy/TAK-102 (minor surgical procedures such as catheter placement are not exclusionary criteria).
13. Previous treatment with any GPC3-targeted therapy.
14. Any unresolved toxicity greater than Grade 2 from previous anticancer therapy.
15. Participants with risk of bleeding as judged by the investigator(s).
16. Presence of central nervous system (CNS) metastasis or other significant neurological conditions (participant with CNS metastases that have been effectively treated where necessary and stable can be enrolled).
17. Participants with medically diagnosed past or current hepatic encephalopathy.
18. Participants with positive human immunodeficiency virus (HIV) and/or human T-cell lymphotrophic virus (HTLV) infection.
19. Participants with clinically significant ascites, which is defined as ascites that are physically positive or require intervention (eg, puncture or medication) for control; those whose imaging result shows ascites requiring no intervention may be included.
20. Participants with a history of organ transplantation or awaiting organ transplantation.
21. Participants with severe immediate hypersensitivity to any of the agents including cyclophosphamide, fludarabine, ganciclovir, or streptomycin.
22. Admission or evidence of illicit drug use, drug abuse, or alcohol abuse.
23. Female participants who are lactating and breastfeeding or have a positive serum pregnancy test (urine pregnancy test is allowed before treatment with preconditioning chemotherapy and TAK-102).

Note: Female participants who are lactating will be eligible if they discontinue breastfeeding before the treatment with TAK-102.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with First Cycle Dose-Limiting Toxicities (DLTs) | Up to 28 days
  Toxicity will be evaluated according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 5.0. DLT will be defined as any of the events specified in the protocol that are considered by the investigator to be at least possibly related to therapy with study medications.
Number of Participants With One or More Treatment-emergent Adverse Event (TEAE) | Up to 3 year
  An adverse event (AE) means any untoward medical occurrence in a participant administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it is related to the medicinal product. This includes any newly occurring event, or a previous condition that has increased in severity or frequency since the administration of study drug.
Number of Participants With Adverse Events of Clinical Interest | Up to 3 year
  Adverse events of clinical interest include severe immune effector cell-associated neurotoxicity syndrome (ICANS), cytokine release syndrome (CRS), hemophagocytic lymphohistiocytosis (HLH), macrophage activation syndrome (MAS), tumor lysis syndrome (TLS), and liver function abnormality.

SECONDARY OUTCOMES:
Objective response based on the investigator's assessment using study-specific modified Response Evaluation Criteria in Solid Tumors Version 1.1 (ssmRECIST 1.1) | Up to 3 year
  Objective Response will be assessed by the investigators with ssmRECIST 1.1 and disease response criteria are following; Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of 1 or more new lesions. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Duration of Response (DOR) as Assessed by the Investigator | Up to 3 year
  DOR is defined as the time from the date of first documentation of a PR or better (determined by the investigator) to the date of first documentation of progressive disease (PD) for responders (PR or better) per RECIST version 1.1, after the initiation of study treatment. Responders without documentation of PD will be censored at the date of last response assessment that is SD or better. CR: Disappearance of all target lesions. PR: At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD. PD: At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of 1 or more new lesions. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Disease Control Rate (DCR) as Assessed by the Investigator | Up to 3 year
  DCR is defined as the percentage of participants who achieve SD or better (determined by the investigator) ≥6 weeks during the study in response-evaluable population per RECIST version 1.1, after the initiation of study treatment. CR: Disappearance of all target lesions. PR: At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD. Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of 1 or more new lesions. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time to Progression as Assessed by the Investigator | Up to 3 year
  TTP is defined as the time from the date of study drug administration to the date of first documented disease progression by the investigator.
Progression-Free Survival (PFS) as Assessed by the Investigator | Up to 3 year
  PFS is defined as the time from the TAK-102 infusion date to the date of disease progression or death from any cause.
Overall Survival (OS) | Up to 3 year
  OS is defined as the time from the TAK-102 infusion to the date of death from any cause.
Maximum (Peak) Observed in Peripheral Blood Product Concentration after Single Dose Administration (Cmax) Evaluated by CAR Copy Number | Up to 3 year; Before-infusion and multiple time points (Day 1,2,5,7,9,11,14,17,21.28, Month 2 to 6 and Month 7-12, 18, 24, 30 and 36) post-dose after the intravenous infusion
Time of First Occurrence of Maximum Observed in Peripheral Blood Concentration (Tmax) Evaluated by CAR Copy Number | Up to 3 year; Before-infusion and multiple time points (Day 1,2,5,7,9,11,14,17,21.28, Month 2 to 6 and Month 7-12, 18, 24, 30 and 36) post-dose after the intravenous infusion
Last Observed Quantifiable Concentration in Peripheral Blood (Clast) Evaluated by CAR Copy Number | Up to 3 year; Before-infusion and multiple time points (Day 1,2,5,7,9,11,14,17,21.28, Month 2 to 6 and Month 7-12, 18, 24, 30 and 36) post-dose after the intravenous infusion
Time of Last Observed Quantifiable Concentration in Peripheral Blood (Tlast) Evaluated by CAR Copy Number | Up to 3 year; Before-infusion and multiple time points (Day 1,2,5,7,9,11,14,17,21.28, Month 2 to 6 and Month 7-12, 18, 24, 30 and 36) post-dose after the intravenous infusion
Area Under the Plasma Concentration-Time Curves (AUCs) Evaluated by CAR Copy Number | Up to 3 year; Before-infusion and multiple time points (Day 1,2,5,7,9,11,14,17,21.28, Month 2 to 6 and Month 7-12, 18, 24, 30 and 36) post-dose after the intravenous infusion
Number of Cases with Replication Competent Retrovirus (RCR)-Positive Test Results | Up to 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (3):
- Japan (3):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Kyoto University Hospital, Kyoto

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be re-identified (due to the limited number of study participants).

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b603d4db2bf003ab4a39f